CLINICAL TRIAL: NCT00047671
Title: Ethnic Variations in Antidepressant Response
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Lisa Glassman, Cedars-Sinai Medical Center, Department of Psychiatry, Clinical Trials Unit
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH062531 (NIH); EVA-00183-02; DATR A5-ETMA
Record Dates: First submitted 2002-10-11; First posted 2002-10-16 (Estimated); Last update posted 2009-08-04 (Estimated); Status verified 2009-08

CONDITIONS: Depression
Keywords: Depressive Disorder
MeSH Terms: conditions — Depression; Depressive Disorder | interventions — Citalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Citalopram (Active Comparator): All subjects receive an FDA approved dose of Citalopram
  Interventions: Drug: Citalopram

INTERVENTIONS:
Drug: Citalopram — PDA Approved antidepressant

SUMMARY:
This 11-week study aims to determine how genetic factors affect the way African Americans and Caucasians with major depression respond to antidepressant medication [citalopram (Celexa®)].

DETAILED DESCRIPTION:
Depressed patients vary substantially in their responses to antidepressants. Genetic factors may account for a large part of these differences in response. This study will include both African Americans and Caucasians to examine the role of genetic factors in treatment response.

Participants receive citalopram (Celexa) for 8 weeks and a placebo for 1 week. Visits occur once a week for 11 weeks. A variety of interviews, scales, tests, and questionnaires are used to assess participants.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV criteria for Major Depression
* African-American or Caucasian ethnic background (both parents and 3 out of 4 grandparents)

Exclusion Criteria:

* Schizophrenia, schizophreniform disorder, schizoaffective disorder, schizotypal disorder, psychotic depression, or bipolar disorder
* Current drug abuse or history of drug abuse within the past 6 months
* Unstable medical or neurological conditions that interfere with the treatment of depression
* Allergy to citalopram
* Failure to respond to adequate citalopram drug trial (40 mg for at least 6 weeks)
* Seizure disorder
* Pregnancy
* Psychotropic medications, including antidepressants and neuroleptics
* Suicidal ideation or other safety issues
* Fluoxetine (Prozac) or MAOIs (Nardil, Parnate) in the last 2 months
* Ongoing cognitive behavioral therapy or intensive psychotherapy. General talk therapy is acceptable

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2002-06; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression | Measured weekly for 11 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Cedars-Sinai Medical Center, Department of Psychiatry, Clinical Trials Unit, Los Angeles, California
  - UCLA/King-Drew, Los Angeles, California
  - Harbor-UCLA Medical Center, Torrance, California

REFERENCES:
- [Derived] Poland RE, Lesser IM, Wan YJ, Gertsik L, Yao J, Raffel LJ, Lin KM, Myers HF. Response to citalopram is not associated with SLC6A4 genotype in African-Americans and Caucasians with major depression. Life Sci. 2013 May 30;92(20-21):967-70. doi: 10.1016/j.lfs.2013.03.009. Epub 2013 Apr 3. PMID 23562852
- [Derived] Joseph NT, Myers HF, Schettino JR, Olmos NT, Bingham-Mira C, Lesser IM, Poland RE. Support and undermining in interpersonal relationships are associated with symptom improvement in a trial of antidepressant medication. Psychiatry. 2011 Fall;74(3):240-54. doi: 10.1521/psyc.2011.74.3.240. PMID 21916630